CLINICAL TRIAL: NCT06334536
Title: Multi-country Survey on Violence Against Women Among Medical Staff.
Status: Not yet recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Asia and Oceania Federation of Obstetrics and Gynaecology (Unknown)
Responsible Party: Principal Investigator, Unnop Jaisamrarn, Professor, Chulalongkorn University
Other Study IDs: 0832/66
Record Dates: First submitted 2024-03-19; First posted 2024-03-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-03

CONDITIONS: Violence Against Women
Keywords: medical staff; violence against women; gender-based violence; knowledge; attitude; practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Medical staff: Medical staff who work at the Department of Obstetrics and Gynecology or Women Health Units in Asia and Oceania countries.

SUMMARY:
The goal of this observational study is to investigate the knowledge, attitude, and practice (KAP) towards violence against women (VAW) among medical staff in the Department of Obstetrics and Gynecology in Asia and Oceania countries

The main question it aims to answer is:

* the KAP towards VAW among medical staff in the Department of Obstetrics and Gynecology in Asia and Oceania countries
* the KAP towards support service of VAW among medical staff in the Department of Obstetrics and Gynecology in Asia and Oceania countries

Participants will be asked to complete the online self-administrated questionnaire.

DETAILED DESCRIPTION:
The medical staff in the Department of Obstetrics and Gynecology or Women Health Units are in an optimal position to address VAW.

This survey aimed to investigate 1) the KAP towards VAW among medical staff in the Department of Obstetrics and Gynecology in Asia and Oceania countries, and 2) KAP towards the support service of VAW among medical staff in the Department of Obstetrics and Gynecology in Asia and Oceania countries.

This multinational, cross-sectional study will be carried out using an online self-administrated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Any medical staff in Department of Obstetrics and Gynecology or Women Health Units, who are aged 18 and over and agree to fill out the questionnaire will be eligible to participate in this study.

Exclusion Criteria:

* There is no demographic restriction on participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any medical staff in the Department of Obstetrics and Gynecology or Women Health Units, who are aged 18 and over, and agree to fill the questionnaire will be eligible to participate in this study. Medical staff are licensed healthcare providers (medical doctors, nursing staff, and others).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
KAP towards VAW | through study completion, an average of 1 year
  Using questionnaire to explore the levels of KAP towards VAW among medical staff
KAP towards support service of VAW | through study completion, an average of 1 year
  Using questionnaire to explore the levels of KAP towards support service of VAW among medical staff

CONTACTS AND LOCATIONS:
Overall Officials: Unnop Jaisamrarn, MD,MHS, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: Undecided
Since this is the multinational survey, we will decide after discussing with investigators of each country.